CLINICAL TRIAL: NCT03724565
Title: Air Quality Check in Gastrointestinal Endoscopy Unit Using Air Quality Monitoring Sensors
Brief Title: Air Quality Check in Gastrointestinal Endoscopy Unit
Status: Completed | Type: Observational
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Chang Seok Bang, Assistant professor of Hallym University College of Medicine, Chuncheon Sacred Heart Hospital
Other Study IDs: bangairquality
Record Dates: First submitted 2018-10-27; First posted 2018-10-30 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Endoscopy, Gastrointestinal
Keywords: endoscopy, gastrointestinal; air pollution, indoor; Respiratory Protective Devices

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Endoscopic procedural area: air quality check of endoscopic procedural room
  Interventions: Procedure: Method of endoscopic procedure
- Recovery area for patients: air quality check of recovery area for patients in endoscopic unit
- Cleansing area for equipments: air quality check of cleansing area for equipments in endoscopic unit

INTERVENTIONS:
Procedure: Method of endoscopic procedure — Air quality according to the method of endoscopic procedure will be checked (for example, upper diagnostic endoscopy, colonoscopy, endoscopic submucosal dissection, endoscopic mucosal resection, etc)
  Groups: Endoscopic procedural area

SUMMARY:
Air pollution sources in indoor area are one of the main factors for reducing indoor air quality of locations. A gastrointestinal endoscopy unit consists of the following area: procedural, recovery areas, and area for a disinfection and cleaning for equipment. This area is frequently exposed to the gastrointestinal gas expelled from patients and gas from electrocoagulated tissue through carbonation or electrocoagulation of neoplasms. This can be potential harmful component for respiratory health not only to medical practitioners but also to the patients who undergo endoscopic examinations. However, there has been scare data for the air quality check in the endoscopic unit.

DETAILED DESCRIPTION:
Air pollution sources in indoor area are one of the main factors for reducing indoor air quality of locations. A gastrointestinal endoscopy unit consists of the following area: procedural, recovery areas, and area for a disinfection and cleaning for equipment. This area is frequently exposed to the gastrointestinal gas expelled from patients and gas from electrocoagulated tissue through carbonation or electrocoagulation of neoplasms (procedure of endoscopic submucosal dissection, endoscopic mucosal resection, etc). This can be potential harmful component for respiratory health not only to medical practitioners but also to the patients who undergo endoscopic examinations. However, there has been scare data for the air quality check in the endoscopic unit. The aim of this study is to check the air quality using conventional portable passive air quality monitoring sensors in gastrointestinal endoscopy unit.

ELIGIBILITY:
Inclusion Criteria:

* This study will check the only air quality in endoscopic unit of Hallym University Chuncheon Sacred Heart hospital of Korea, not a patients.

Exclusion Criteria:

* This study will check the only air quality in endoscopic unit of Hallym University Chuncheon Sacred Heart hospital of Korea, not a patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will check the only air quality in endoscopic unit of Hallym University Chuncheon Sacred Heart hospital of Korea, not a patients.
Sampling Method: Non-Probability Sample
Enrollment: 4320 (Actual)
Dates: Start 2018-06-17 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
atmospheric Carbon dioxide (CO2) | up to 1 week
  CO2 ppb level in the area of endoscopic unit
atmospheric total volatile organic compound (TVOC) | up to 1 week
  TVOC ppb level in the area of endoscopic unit
atmospheric particulate matter that have a diameter of less than 2.5 micrometer (PM2.5) | up to 1 week
  PM2.5 ug/m3 level in the area of endoscopic unit
atmospheric nitrogen dioxide (NO2) | up to 1 week
  NO2 ppb level in the area of endoscopic unit
atmospheric carbon mono-oxide (CO) | up to 1 week
  CO ppb level in the area of endoscopic unit
atmospheric ozone | up to 1 week
  ozone ppb level in the area of endoscopic unit

SECONDARY OUTCOMES:
atmospheric temperature | up to 1 week
  atmospheric temperature in the area of endoscopic unit
atmospheric humidity | up to 1 week
  atmospheric humidity in the area of endoscopic unit
atmospheric pressure | up to 1 week
  atmospheric pressure in the area of endoscopic unit

CONTACTS AND LOCATIONS:
Overall Officials: Chang Seok Bang, MD, PhD, Principal Investigator — Hallym University College of Medicine, Korea
Locations (1):
- Chuncheon Sacred Heart hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There will be no patients-related data in this study (ecologic study)

REFERENCES:
- [Derived] Bang CS, Lee K, Yang YJ, Baik GH. Ambient air pollution in gastrointestinal endoscopy unit. Surg Endosc. 2020 Sep;34(9):3795-3804. doi: 10.1007/s00464-019-07144-8. Epub 2019 Oct 3. PMID 31583470